CLINICAL TRIAL: NCT03786107
Title: HER-Seq: A Blood-based Screening Study to Identify Patients With HER2 Mutations for Enrollment Into Clinical Research Studies of Neratinib
Status: Terminated | Type: Observational
Why Stopped: The study was stopped early due to increased global access to genomic screening. It is no longer economical to continue with this particular single-gene screening protocol.
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PUMA-NER-9501
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Hormone Receptor-Positive, HER2-Negative Metastatic Breast Cancer; Metastatic Cervical Cancer
Keywords: Circulating Tumor DNA; HER2; Genomic Screening; Metastatic; Breast; Cervical; ERBB2; Mutation; CDK4/6; HR Positive
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating tumor DNA from plasma will be collected from eligible participants. ERBB2 (HER2) gene exons 8 and 17-24 will be sequenced by next generation sequencing (NGS) at a central laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Diagnostic Test: Almac HER-Seq Assay — whole blood sample analysis

SUMMARY:
This is a multi-center, observational genomic screening protocol to identify participants whose tumors harbor somatic mutations in the ERBB2 (HER2) gene, as measured in circulating tumor DNA (ctDNA) . Participants with histologically confirmed, hormone receptor positive, HER-2 negative, metastatic breast cancer (MBC) or metastatic cervical cancer (MCC) are eligible for screening at 6 months intervals, or if disease progression is suspected/confirmed. Blood samples will be collected from eligible participants and ctDNA will be extracted and sequenced at a central laboratory, using a HER2-targeted next generation sequencing (NGS) test. A certified molecular test report will be issued from the central laboratory and provided to the investigators and the study sponsor. Participants who are identified with HER2 mutations by this screening protocol will subsequently have access to an appropriate neratinib treatment protocol, pending medical eligibility.

ELIGIBILITY:
Inclusion Criteria:

* Women and men who are ≥18 years old at signing of informed consent
* Eastern Cooperative Oncology Group (ECOG) status of 0 to 2
* Provide written informed consent to participate in the study and for circulating tumor DNA screening
* Must be able to provide blood sample(s) for HER2 mutation testing
* Participants with imaging or histologically confirmed, HR-positive, HER2-negative MBC who are presently receiving or have received CDK4/6 inhibitor as a prior therapy in any setting, or participants with imaging or histologically confirmed metastatic cervical cancer
* At least one measurable lesion, as defined by RECIST v1.1

Exclusion Criteria:

* Participants with breast cancer with known HER2-positive or HER2-amplified tumors
* Participants with breast cancer with HR-negative tumors
* Participants who have received HER2-directed TKI
* Participants with previously documented somatic KRAS activating mutation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with histologically-confirmed metastatic breast or metastatic cervical cancer
Sampling Method: Non-Probability Sample
Enrollment: 1583 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants Eligible for Neratinib Treatment | From enrollment date to identification of HER2 positive mutation, assessed up to five years
  Identification of participants with somatic, activating HER2 mutations who might qualify for enrollment into neratinib treatment protocols

CONTACTS AND LOCATIONS:
Overall Officials: Senior Vice President Clinical Science and Pharmacology, Study Director — Puma Biotechnology, Inc.
Locations (22):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States
- Institut Curie, Saint-Cloud, France
- Ireland (5):
  - Cork University Hospital, Wilton, Cork
  - St. Vincent's University Hospital, Elm Park, Dublin
  - Mater Misericordiae University Hospital, Institute for Cancer Research, Dublin
  - Beaumont Hospital, Cancer Clinical Trials & Research Unit, Dublin
  - University Hospital Waterford, Department of Medical Oncology, Waterford
- Israel (4):
  - Rabin Medical Center, Davidoff Cancer Center, Petah Tikva, Central District
  - Kaplan Medical Center, Rehovot, Central District
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli, Italy
- Institute for Oncology and Radiology of Serbia, Belgrade, Serbia
- Spain (9):
  - Hospital Universitario Quirónsalud Madrid, Pozuelo de Alarcón, Madrid
  - Instituto Oncológico Dr. Rosell, Hospital Universitario Quirón Dexeus, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - START Madrid, Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Fundación Instituto Valenciano de Oncológia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Puma Biotechnology is committed to sharing clinical trial data and information to help physicians and patients make informed treatment decisions, and to help qualified researchers advance scientific knowledge.
  In accordance with legal and regulatory requirements, Puma publishes study protocol information and clinical study results on clinical trial registries, including ClinicalTrials.gov and EU Clinical Trials Register. Puma also publishes information about clinical studies in peer-reviewed scientific journals and shares data in scientific meetings.
  Puma commits to safeguarding confidentiality and patient privacy throughout the clinical trial data and information sharing process. Any patient-level data will be anonymized to protect personally identifiable information.
  Qualified researchers and study participants may submit requests for other study documentation and clinical trial data to clinicaltrials@pumabiotechnology.com for consideration.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Clinical study documents and clinical trial data may be requested by qualified researchers and study participants for studies that have been completed for at least 18 months, and for which the indication of the drug has been approved in the US and/or EU, as applicable. Requests will be accepted for up to 24 months after the criteria described in this section are met.
Access Criteria: Requestors must provide organizational contact information; a detailed research plan, including outcomes; timeline for completion of the research; qualifications of the research team; funding source; and potential conflicts of interest.
  Puma will not provide access to patient-level data if there is a reasonable likelihood that individual patients could be identified, or in cases where confidentiality or consent provisions prohibit transfer of data or information to third parties. Additionally, Puma will not disclose information that jeopardizes intellectual property rights or divulges confidential commercial information.
URL: https://pumabiotechnology.com/data_sharing_policy.html